CLINICAL TRIAL: NCT06130891
Title: Effects of Cognitive Exercises With Sensory Motor Relearning Program on Upper Limb Function in Sub-Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/ 0244 Hifsa Waheed
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Ischemic
Keywords: cognitive exercise therapy; sensory motor relearning; upper limb function
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive sensory motor relearning Group (Experimental): Cognitive, sensory, and motor training
  Interventions: Other: Cognitive sensory motor relearning
- Sensory Motor Relearning Group (Experimental): Sensory and motor training
  Interventions: Other: Sensory motor relearning
- Motor Relearning Group (Experimental): Motor training
  Interventions: Other: Motor Relearning

INTERVENTIONS:
Other: Cognitive sensory motor relearning — Cognitive Exercises:
  * Orientation: Checking awareness of date, time, and weather.
  * Attention: Tasks like connecting dots or spotting differences.
  * Shape Sorting: Sorting objects by size, color, etc.
  * Calculation Training: Counting money, beads, basic arithmetic.
  * Memory: Recalling objects on a tray, numbers backward, word associations.
  Sensory Relearning:
  * Discrimination: Identifying textures, shapes, sizes, and temperatures.
  * Tactile Recognition: Recognizing objects through touch.
  * Proprioception: Matching affected limb's position to unaffected limb's.
  Motor Relearning:
  * Task-Specific Training: Grasping, pouring, wiping, screwing, holding objects.
  * Progression: Increasing duration, intensity, and resistance. 45 minutes per day, 5 days a week for 6 weeks.
  Arms: Cognitive sensory motor relearning Group
Other: Sensory motor relearning — Sensory Relearning:
  * Discrimination: Identifying textures, shapes, sizes, and temperatures.
  * Tactile Recognition: Recognizing objects through touch.
  * Proprioception: Matching affected limb's position to unaffected limb's.
  Motor Relearning:
  * Task-Specific Training: Grasping, pouring, wiping, screwing, holding objects.
  * Progression: Increasing duration, intensity, and resistance. 45 minutes per day, 5 days a week for 6 weeks.
  Arms: Sensory Motor Relearning Group
Other: Motor Relearning — Motor Relearning:
  * Task-Specific Training: Grasping, pouring, wiping, screwing, holding objects.
  * Progression: Increasing duration, intensity, and resistance. 45 minutes per day, 5 days a week for 6 weeks.
  Arms: Motor Relearning Group

SUMMARY:
The goal of this clinical trial is to compare the effects of cognitive sensory motor relearning, and sensory-motor relearning program alone on manual ability, sensation, gross and fine movements, and cognition in post-stroke patients. The main aim is to evaluate the effectiveness of an integrated approach and its impact on motor function, sensory processing, and cognitive skills in sub-acute stroke patients, with the goal of contributing to the development of more efficient rehabilitation interventions for UL sensory-motor impairments after stroke.

DETAILED DESCRIPTION:
Stroke is not only associated with a high mortality rate, but It also leads to major disabilities. The American Heart Association reported that nearly 75% of stroke victims have dysfunction and 15-30% of stroke survivors have severe disability. Stroke survivors often suffer from impaired motor function, sensory processing, and cognitive abilities depending on the severity and site of the lesion, severely impacting their functional independence and quality of life. About 80% of stroke survivors experience some degree of impairment in their UL which includes loss of dexterity, abnormal muscle tone, loss of coordinated movements, and diminished sensations depending upon to nature of the lesion.

Cognitive exercise treatment is a motor learning model that focuses on high-level cognitive function and occurs through the integration of perception-cognition-activity processes, such as motor regulation. Activation of the brain's cognitive process, which includes perception, memory, attention, language, and decision-making, is the core of cognitive training. Most studies have focused on either sensory, motor, or cognitive interventions separately, overlooking the potential benefits of simultaneously addressing these domains. This combined intervention targets not only motor skills, but also cognitive skills, sensory processing, and manual dexterity. By addressing physical and cognitive domains simultaneously, this study aims to evaluate the effectiveness of an integrated approach and its impact on motor function, sensory processing, and cognitive skills in sub-acute ischemic stroke patients, with the goal of contributing to the development of more efficient rehabilitation interventions for UL sensory-motor impairments after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients.
* 45- 60 years of age.
* 1st ever stroke.
* Sub-acute ischemic stroke.
* 8-12 weeks post stroke patients.
* Participants must have motor and somatosensory deficits in the upper limb on the affected side, as indicated by an ARAT score between 40 and 50 out of 57.
* Participants must be able to provide informed consent or have a legal representative who can provide informed consent on their behalf.
* MoCA score between 18-24
* Modified Ashworth scale < +1

Exclusion Criteria:

* Participants who have a history of significant neurological or psychiatric disorders, other than stroke, that could interfere with upper limb motor or sensory recovery.
* Participants who have other medical conditions that could interfere with therapy or assessments, such as severe arthritis or joint injuries.
* Participants who have severe visual or hearing impairments that would interfere with therapy or assessments.
* Participants who are currently participating in another clinical trial or research study.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | 6 weeks
  Changes from baseline The instrument contains 19 items grouped into 4 sub-tests: grasp, grip, pinch, and gross motor. Item performance is rated on a 4-point scale (0=unable; 1=partial; 2= abnormal; 3=normal) then item ratings are summed and reported out of 57 points with higher score indicating greater UE function.
Revised Nottingham Sensory Assessment (Somatosensory Impairments) | 6 weeks
  Changes from baseline rNSA examines somatosensory impairment using a 3-point scale (0 =absent, 1 = impaired, 2 = normal) and takes approximately 25-35 min to complete. It consists of 72 items grouped into three sub-scales measuring tactile sensation, proprioception, and stereognosis. The Tactile Sensation subscale includes light touch, temperature, pinprick, pressure, tactile localization, and bilateral simultaneous touch. Higher scores demonstrate better somatosensory function.
ABILHAND questionnaire (ABIL) | 6 weeks
  Changes from baseline ABILHAND is an inventory of 23 manual activities that the patient is originally asked to judge on a 3-level scale: 0 (impossible), 1 (difficult), and 2 (easy). The test explores bi-manual activities done without other human or technical help. For each question the patient provided his/her feeling of difficulty irrespective of the limb(s) actually used to do the activity. Activities not attempted in the last 3 months are not scored and encoded as missing responses.
MoCA (Montreal Cognitive Assessment) | 6 weeks
  Changes from baseline Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- THQ Hospital, Muridke, Sheikhupura, Punjab, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No